CLINICAL TRIAL: NCT00427531
Title: An Exploratory Trial to Examine the Accuracy of Various Hot Flash Variables With an Ambulatory Sternal Skin Conductance Recording Tool
Brief Title: Skin Conduction Device and Patient Diary for Measuring Hot Flashes in Postmenopausal Women With Hot Flashes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Debra L. Barton, R.N., Ph.D., Mayo Clinic Cancer Center
Purpose: Diagnostic
Other Study IDs: CDR0000525737; P30CA015083 (NIH); MC06C3 (Other: Mayo Clinic Cancer Center); 06-002452 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Last update posted 2011-03-17 (Estimated); Status verified 2011-03

CONDITIONS: Hot Flashes
Keywords: hot flashes
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: physiologic testing

SUMMARY:
RATIONALE: Measuring how often hot flashes occur in postmenopausal women may be done by using a skin conduction device or by using a diary.

PURPOSE: This clinical trial is studying a skin conduction device and a patient diary for measuring hot flashes in postmenopausal women with hot flashes.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the differences in frequency, severity, and duration of hot flash activity using an ambulatory sternal skin conductance recording tool and patient hot flash diary in postmenopausal women with hot flashes.
* Assess the recordings made by an ambulatory sternal skin conductance measuring and recording tool during a 30-minute exercise period in these patients.

OUTLINE: Patients wear an ambulatory sternal skin conductance hot flash device continuously for 24 hours.

Patients complete hot flash diaries over 24 hours. Patients undergo treadmill exercise over 30 minutes and record hot flash activity using the skin conductance device during 10 minutes of sweating. Patients also complete the Comfort, Bother, and Weight Questionnaire at the completion of the study.

PROJECTED ACCRUAL: A total of 3 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of bothersome hot flashes, defined by their occurrence ≥ 4 times/day

  * Daily hot flashes that have been present for ≥ 1 month

PATIENT CHARACTERISTICS:

* Female
* Postmenopausal
* ECOG performance status 0-1
* No history of allergic or other adverse reactions to adhesives
* No other medical condition known to cause sweating and/or flushing
* No implanted pacemakers or metal implants
* No reliance on electronic devices for regular monitoring (i.e., insulin pumps or blood pressure monitors)

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2006-06; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Differences in frequency, severity, and duration of hot flash activity using an ambulatory sternal skin conductance recording tool and patient hot flash diary
Hot flash recordings as measured by an ambulatory sternal skin conductance measuring and recording tool during a 30-minute exercise period

CONTACTS AND LOCATIONS:
Overall Officials: Debra L. Barton, R.N., Ph.D., Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States